CLINICAL TRIAL: NCT00180635
Title: A Double Blind, Crossover Placebo-controlled Study to Evaluate the Effect of L-arginine and Aminoguanidine on Bronchial and Alveolar Nitric Oxide and Nitric Oxide Metabolites
Brief Title: NO Donors and Inhibitors to Study Imbalance of Nitrogen Stress and Antioxidant Defense in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02-104-170903
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Aminoguanidine; Nitric oxide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — pimagedine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Healthy volunteers non smoker (Experimental): Control group
  Interventions: Drug: Aminoguanidine; Drug: Placebos
- Healthy volunteers smoker (Experimental): More than 10 pack-years
  Interventions: Drug: Aminoguanidine; Drug: Placebos
- Chronic Obstructive Pulmonary Disease COPD (Experimental): COPD diagnosed according to the Global Initiative for Chronic Obstructive Lung Disease guidelines
  Interventions: Drug: Aminoguanidine; Drug: Placebos

INTERVENTIONS:
Drug: Aminoguanidine — 500mg
  Other Names: Nebulased Aminoguanidine
Drug: Placebos — 2ml
  Other Names: Nebulase saline solution

SUMMARY:
The primary aim of this study is to investigate the effects of oral and inhaled administration of L-arginine and of inhaled aminoguanidine on bronchial and alveolar exhaled NO and NO metabolites in exhaled breath condensate, induced sputum, nasal lavage and mouth wash fluid in healthy non-smokers, current smokers and patients with COPD.

DETAILED DESCRIPTION:
Nitric oxide (NO) is produced by resident and inflammatory cells in the respiratory tract by the enzyme NO synthase (NOS), which exists in three isoforms: neuronal NOS (nNOS), inducible NOS (iNOS), and endothelial NOS. NO production is increased in patients with COPD, and the production of NO under oxidative stress conditions generates reactive nitrogen species that may amplify the inflammatory response in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smokers
* Normal spirometry (FEV1 >90 % predicted; exhaled NO bigger than or equal to 10 ppb; flow 50 ml/s)
* At risk (current smokers)

  * Normal spirometry, with or without chronic symptoms (cough, sputum production)
  * FEV1 reversibility of <15% after inhaled beta2-agonists*
* Moderate COPD

  * FEV1 greater than or equal to 30% and < 80%
  * FEV1/FVC < 70% predicted
  * FEV1 reversibility of <15% after inhaled beta2-agonists
  * With or without chronic symptoms (cough, sputum production, dyspnea)
* Able to comprehend and grant a written informed consent

Exclusion Criteria:

* Concomitant use or pre-treatment within the last 4 weeks with oral steroids
* Respiratory infection within 4 weeks prior to entry into the trial
* Females who are pregnant or lactating
* History of current or past drug or alcohol abuse

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-10 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Bronchial exhale nitric oxide (JNO) | 24 hours
  Bronchial exhale nitric oxide (JNO) as assessed by Chemo luminescence

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brindicci C, Ito K, Torre O, Barnes PJ, Kharitonov SA. Effects of aminoguanidine, an inhibitor of inducible nitric oxide synthase, on nitric oxide production and its metabolites in healthy control subjects, healthy smokers, and COPD patients. Chest. 2009 Feb;135(2):353-367. doi: 10.1378/chest.08-0964. Epub 2008 Aug 21. PMID 18719059